CLINICAL TRIAL: NCT01410565
Title: A Phase 3 International, Multicenter, Double-Blind, Placebo-Controlled, Randomized Trial Evaluating the Efficacy and Safety of Multiple Instillations of Intravesical Apaziquone vs. Placebo in Patients With Low-Intermediate Risk Non-Muscle Invasive Bladder Cancer (NMIBC)
Brief Title: Efficacy and Safety of Multi-Instillations of Apaziquone in Patients With Non-Muscle Invasive Bladder Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business reason
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPI-1011
Record Dates: First submitted 2011-08-01; First posted 2011-08-05 (Estimated); Results first posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Non-Muscle Invasive Bladder Cancer; NMIBC; Apaziquone; EOquin; GU Cancer; TURBT
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — apaziquone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apaziquone (Active Comparator)
  Interventions: Drug: Apaziquone
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apaziquone — Apaziquone 4 mg in 40 mL diluent
  Other Names: EO9; EOquin
  Arms: Apaziquone
Drug: Placebo — Placebo for Double Blind Phase
  Arms: Placebo

SUMMARY:
This is an international, multicenter, double-blind, placebo-controlled, randomized study. All eligible patients entering the open label phase of the study will receive a single immediate instillation of apaziquone (4 mg in 40 mL diluent), post transurethral resection-bladder tumor (TURBT). Following Central Pathology review of histology and Double Blind Phase qualification, patients with confirmed eligibility will be randomized to receive either 6 weekly intravesical instillations of apaziquone or matching placebo and undergo cystoscopic and safety assessments every 3 months for 24 months from randomization. Patients with histologic evidence of recurrent disease during the study will be treated according to current treatment guidelines or local standard of care. Safety and efficacy assessments will be performed at 3 month intervals for all randomized patients throughout the study. Patients who receive single dose of apaziquone immediately following TURBT and are not eligible for randomization will be followed for 3 months by cystoscopic exam and safety assessments.

ELIGIBILITY:
Inclusion Criteria:

Open Phase Inclusion Criteria:

1. Has the patient given written informed consent and is the patient willing and able to abide by the protocol?
2. Is the patient 18 years old or above?
3. If the patient is a female of childbearing potential, is she using an acceptable/effective method of contraception?
4. Does the female patient of childbearing potential have a negative serum pregnancy test at screening?
5. Does the patient with clinically apparent primary or recurrent low grade Ta NMIBC have :

   * multiple tumors (2-7)
   * No single Tumor > 3 cm
   * No history / evidence of Tis

   Or does the patient with clinically apparent primary or recurrent high grade Ta NMIBC have:
   * A single tumor that is ≤ 3 cm
   * No history / evidence of Tis
6. Is the patient able to retain bladder instillations for a minimum of 60 minutes?
7. Did the patient have upper urinary tract evaluation to exclude urothelial carcinoma, hydronephrosis or renal cell carcinoma or other renal cancers in the 6 months prior to study screening?
8. Is patient's urethra (including prostatic urethra in men) endoscopically free of any visible TCC?
9. For patients with recurrent tumor, did the patient have at least a 6-month cystoscopically-confirmed tumor-free interval between the last tumor recurrence and the time of screening?
10. Has the male patient with a prostate specific antigen (PSA) between 4 and 10 ng/mL had a diagnostic evaluation that reasonably excludes the diagnosis of prostate cancer in the opinion of the Investigator?

Double-Blind Phase Inclusion Criteria:

1. Was all visible tumor resected at the initial TURBT?
2. Does Central Pathology review of the patient's bladder tumor confirm:

   * Low grade Ta disease for multiple tumors (2 - 7) or
   * High Grade Ta disease for single tumor
   * No microscopic evidence of lymphovascular invasion and/or evidence of tumor thromboemboli

Exclusion Criteria:

Open Phase Exclusion Criteria:

1. Has the patient received any previous pelvic radiotherapy (includes external beam and/or brachytherapy)?
2. Has the patient ever received apaziquone?
3. Has the patient received an induction course (completed 5 of 6 scheduled weekly instillations) of intravesical BCG (± interferon) with the last dose given less than 12 months ago?
4. Has the patient had any prior intravesical chemotherapy, exclusive of single-dose adjuvant intravesical chemotherapy immediately post-TURBT?
5. Does the patient have a history of urinary retention or a post void residual ≥ 250 cc by bladder scan or ultrasound (post void residual test may be repeated up to 3 times)?
6. Does the patient have or has the patient had any bladder tumor with histology other than transitional cell carcinoma?
7. Does the patient have or has the patient had micro-papillary transitional cell carcinoma?
8. If the patient has recurrent papillary disease of the bladder, has the pathology been anything other than pTa in the past?
9. Does the patient have an active urinary tract infection confirmed by culture or a documented history of recurrent UTI (≥ 6 for females and ≥2 for males per year) in the prior 2 years?
10. Does the patient have a bleeding disorder or a screening platelet count < 50 x 109/L?
11. Does the patient have a screening hemoglobin < 10 mg/dL?
12. Does the male patient have a serum PSA > 10 ng/mL?
13. Does the patient have a history of Acquired Immunodeficiency Syndrome or HIV positive?
14. Does the patient have a condition or a concurrent severe and/or uncontrolled medical or psychiatric disease (e.g., uncontrolled diabetes, decompensated congestive heart failure, myocardial infarction within 6 months of study, unstable and uncontrolled hypertension, or an active uncontrolled infection), which could compromise participation, compliance with scheduled visits and/or completion of the study?
15. Has the patient participated in an investigational protocol within the past 90 days?
16. Is the patient pregnant or breast feeding?
17. Does the patient have a life expectancy of <3 years?
18. Has the patient had any other malignancy or received therapy for any malignancy in the last five years except

    * non-melanoma skin tumors
    * stage 0 (in situ) cervical carcinoma
    * undetectable PSA for ≥1 year following definitive therapy for localized prostate cancer?
19. Does the patient have documented vesicoureteral reflux or an indwelling ureteral stent?
20. Does the patient have tumor in a bladder diverticulum?
21. Does the patient have a known allergy to red color food dye?

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Show-Li Sun, MD, Study Director — Spectrum Pharmaceuticals, Inc
Locations (47):
- United States (28):
  - Valley Urologic Associates, Glendale, Arizona
  - Precision Trials, LLC, Phoenix, Arizona
  - South Orange County Medical Research Center, Laguna Woods, California
  - The Urology Center of Colorado, Denver, Colorado
  - Connecticut Clinical Research Center, Middlebury, Connecticut
  - Urology Enterprises, Marietta, Georgia
  - North Idaho Urology, Coeur d'Alene, Idaho
  - Idaho Urologic Institute, P.A., Meridian, Idaho
  - Northeast Indiana Research, LLC, Fort Wayne, Indiana
  - First Urology, PSC, Jeffersonville, Indiana
  - Regional Urology, LLC, Shreveport, Louisiana
  - Anne Arundel Urology, Annapolis, Maryland
  - Spectrum Health Medical Group, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Five Valleys Urology, Missoula, Montana
  - Delaware Valley Urology, LLC - Voorhees, Voorhees Township, New Jersey
  - Delaware Valley Urology, LLC-Westampton, Woodlane, New Jersey
  - University Urology Associates, New York, New York
  - Urology Associates of Rochester, LLC, Rochester, New York
  - TriState Urologic Services PSC, Inc., Cincinnati, Ohio
  - Urologic Consultants of Southeastern Pennsylvania, LLP, Bala-Cynwyd, Pennsylvania
  - Urology Health Specialists, Bryn Mawr, Pennsylvania
  - Urological Associates of Lancaster, Lancaster, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates of South Texas, McAllen, Texas
  - Urology of Virginia, PC, Virginia Beach, Virginia
  - Urology of Virginia, PLLC, Virginia Beach, Virginia
  - Integrity Medical Research, LLC, Mountlake Terrace, Washington
- Canada (19):
  - G. Steinhoff Clinical Research Pacific Urologic Research, Victoria, British Columbia
  - Queen Elizabeth II Health Science Center, Halifax, Nova Scotia
  - The Male/Female Health and Research Centre - Royal Court Medical Centre, Barrie, Ontario
  - Brantford Urology Research, Brantford, Ontario
  - G. Kenneth Jansz Medicine Professional Corporation, Burlington, Ontario
  - Urology Resource Centre, Burlington, Ontario
  - Kingston General Hospital / Queen's University, Kingston, Ontario
  - Urology Associates, Urologic Medical Research, Kitchener, Ontario
  - Mor Urology, Inc., Newmarket, Ontario
  - Office of Bernard Goldfarb, North Bay, Ontario
  - Stanley Flax Medical Professional Corporation, North York, Ontario
  - The Fe/Male Health Centre, Oakville, Ontario
  - Urotec, Oshawa, Ontario
  - Urology/Male Infertility, Scarborough Village, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network Princess Margaret Hospital, Toronto, Ontario
  - Centre universitaire de sante McGill, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec

REFERENCES:
- [Background] Cai T, Nesi G, Tinacci G, Zini E, Mondaini N, Boddi V, Mazzoli S, Bartoletti R. Can early single dose instillation of epirubicin improve bacillus Calmette-Guerin efficacy in patients with nonmuscle invasive high risk bladder cancer? Results from a prospective, randomized, double-blind controlled study. J Urol. 2008 Jul;180(1):110-5. doi: 10.1016/j.juro.2008.03.038. Epub 2008 May 15. PMID 18485394
- [Background] Schellens JH, Planting AS, van Acker BA, Loos WJ, de Boer-Dennert M, van der Burg ME, Koier I, Krediet RT, Stoter G, Verweij J. Phase I and pharmacologic study of the novel indoloquinone bioreductive alkylating cytotoxic drug E09. J Natl Cancer Inst. 1994 Jun 15;86(12):906-12. doi: 10.1093/jnci/86.12.906. PMID 8196081
- [Background] Stenzl A, Hennenlotter J, Schilling D. Can we still afford bladder cancer? Curr Opin Urol. 2008 Sep;18(5):488-92. doi: 10.1097/MOU.0b013e32830b8925. PMID 18670272

RESULTS

PARTICIPANT FLOW:
Groups:
- Apaziquone: Apaziquone: Apaziquone 4 mg in 40 mL diluent
  Apaziquone: Apaziquone in the Double Blind Phase
- Placebo: Placebo
  Placebo: Placebo in the Double Blind Phase
Period: Open Label Phase Apaziquone
Arm/Group | Apaziquone | Placebo | Open Label-Apaziquone
Started | 0 | 0 | 66
Completed | 0 | 0 | 58
Not Completed | 0 | 0 | 8
Period: Double Blind Phase
Arm/Group | Apaziquone | Placebo | Open Label-Apaziquone
Started | 13 (All 66 patients received one dose of Apaziquone in the open label phase.) | 15 | 0
Completed | 0 | 0 | 0
Not Completed | 13 | 15 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Population included all randomized patients in the double blind phase.
Groups:
- Apaziquone: Apaziquone 4 mg in 40 mL diluent
  Apaziquone in the Double Blind Phase
- Placebo: Placebo
  Placebo in the Double Blind Phase
- Total: Total of all reporting groups
Arm/Group | Apaziquone | Placebo | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 6 | 9 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (11.77) | 70.5 (12.66) | 68.2 (12.30)
Gender [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 11 | 13 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 13 | 13 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 15 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Recurrence
Description: Time to recurrence is the time from randomization to the date of first histologically confirmed recurrence of bladder cancer (for eligible patients with Low- intermediate risk NMIBC, who had undergone TURBT followed by, a single instillation of apaziquone immediately post TURBT and multiple instillations of apaziquone or placebo).
Time Frame: Recurrence of cancer in the bladder during 24 months of follow-up
Population: All patients who received Apaziquone in the Open Label Phase and subsequently randomized to one of the treatment arms in the Double Blind Phase. Participants without recurrence were censored.
Measure: Mean (Full Range); unit: months
Groups:
- Apaziquone: Apaziquone: Apaziquone 4 mg in 40 mL diluent
  Apaziquone in the Double Blind Phase
Arm/Group | Apaziquone | Placebo
Number analyzed (Participants) | 13 | 15
months | 9.2 [9.2 to 9.2] | 7.3 [2.3 to 8.5]

2. Secondary Outcome: Recurrence Rate at 24 Months
Description: Measurement the number of participants with the recurrence at 24 months.
Time Frame: 24 months
Population: All patients who received Apaziquone in the Open Label Phase and subsequently randomized to one of the treatment arms in the Double Blind Phase.
Measure: Number; unit: participants
Arm/Group | Apaziquone | Placebo
Number analyzed (Participants) | 13 | 15
participants | 1 | 4

3. Secondary Outcome: Participants With Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs will be mainly characterized by the number of treatment emergent adverse events and treatment related AEs that occur or worsen after the first dose of study treatment.
Time Frame: 24 Months from Randomization
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Apaziquone | Placebo
Number analyzed (Participants) | 13 | 15
participants | 11 | 12

ADVERSE EVENTS:
Arm/Group | Apaziquone | Placebo
Serious Adverse Events (participants affected / at risk) | 1/13 | 1/15
Other Adverse Events (participants affected / at risk) | 11/13 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apaziquone (N=13) | Placebo (N=15)
Arterio Sclerosis (Cardiac disorders) | 1 (1) | 0 (0)
Prostate Cancer (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apaziquone (N=13) | Placebo (N=15)
Dysuria (Renal and urinary disorders) | 5 (5) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 4 (4) | 1 (1)
Bladder pain (Renal and urinary disorders) | 2 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 4 (4)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4)
Urinary retention (Renal and urinary disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No